CLINICAL TRIAL: NCT00575367
Title: A Single-Center, Open-Label, Randomized Study of the Pharmacokinetics of AzaSite Ophthalmic Solution Versus Vigamox in the Tears of Healthy Volunteers Following a Single Ocular Administration
Brief Title: Study of AzaSite Versus Vigamox in the Tears of Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Karen Kuhn, Inspire Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 041-101; P08653
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2009-09-17 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Bacterial Infections; Eye Infections
MeSH Terms: conditions — Bacterial Infections; Eye Infections | interventions — Azithromycin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AzaSite (Active Comparator)
  Interventions: Drug: AzaSite (azithromycin ophthalmic solution)
- Vigamox (Active Comparator)
  Interventions: Drug: Vigamox (moxifloxacin hydrochloride ophthalmic solution)

INTERVENTIONS:
Drug: AzaSite (azithromycin ophthalmic solution) — One drop ophthalmic solution at Visit 2
  Arms: AzaSite
Drug: Vigamox (moxifloxacin hydrochloride ophthalmic solution) — One drop ophthalmic solution at Visit 2
  Arms: Vigamox

SUMMARY:
The purpose of this study is to evaluate the drug concentrations of AzaSite compared to Vigamox in tears of healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Have visual acuity, using corrective lenses (no contact lenses) if necessary, in both eyes of at least +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study.
* Have normal lid anatomy.

Exclusion Criteria:

* Have an abnormal biomicroscopy or ophthalmoscopy exam.
* Have a diagnosis of dry eye disease or have experienced any of the dry eye symptoms (photophobia, foreign body sensation, itching, burning, pain, dry or grittiness) in the past thirty days.
* Have used artificial tears in the past thirty days.
* Have a diagnosis of on-going ocular infection or lid margin inflammation.
* Have ever had penetrating ocular surface or intraocular surgery.
* Have a known hypersensitivity to azithromycin, or any macrolide antibiotic or to any of the ingredients in AzaSite.
* Have had a known hypersensitivity to Vigamox or any fluoroquinolone antibiotics or to any of the ingredients in Vigamox.
* Have had corneal or lid abnormalities.
* Have glaucoma, or Intra Ocular Pressure of 22 mm Hg or greater in one or both eyes.
* Have any ocular pathology with the exception of cataracts.
* Have a serious systemic disease or uncontrolled medical condition.
* Have experienced symptoms of viral or allergic conjunctivitis in the past 30 days.
* Have a history of liver or kidney disease resulting in persisting dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AzaSite | Vigamox
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AzaSite | Vigamox | Total
Number analyzed (Participants) | 18 | 17 | 35
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures for two subjects were not included in this analysis due to missing data on too many data points. Although the total number of baseline participants was 37, the actual number included in the analysis was 35 subjects, 18 subjects in the Azasite group and 17 in the Vigamox group.
  years | 33.9 (12.59) | 38.1 (13.29) | 36.0 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Concentration of AzaSite and Vigamox in the Tear Fluid Across Six Time Points Ranging From 15 Minutes to 24 Hours Following Administration.
Time Frame: 15 minutes, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | AzaSite | Vigamox
Number analyzed (Participants) | 18 | 17
µg/mL
  15 Minutes | 16.485 (22.9971) | 8.199 (15.9873)
  1 Hour | 4.007 (4.3680) | 2.221 (4.1506)
  2 Hours | 1.966 (3.6632) | 2.985 (5.6350)
  4 Hours | 1.558 (2.6151) | 0.603 (1.0074)
  8 Hours | 2.590 (4.8111) | 1.364 (2.7629)
  24 Hours | 0.195 (0.2558) | 0.021 (0.0449)

ADVERSE EVENTS:
Arm/Group | AzaSite | Vigamox
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish or discuss trial results until written communication is received from Inspire Pharmaceuticals, Inc.